CLINICAL TRIAL: NCT03946319
Title: A Personalized, Transdiagnostic Approach to Preventative Mental Health Using Machine Learning
Brief Title: Personalized, Transdiagnostic Approach to Preventative Mental Health
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Introspect Health (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: IH-001
Record Dates: First submitted 2019-05-08; First posted 2019-05-10 (Actual); Last update posted 2019-05-14 (Actual); Status verified 2019-05

CONDITIONS: Mental Health; Mental Disorders; Delivery of Health Care; Self-Assessment; Diagnosis, Psychiatric
Keywords: Internet Interventions; eMental Health; mHealth; Transdiagnostic; Behavioral Health; Wellness; Connected Health; Introspect
MeSH Terms: conditions — Psychological Well-Being; Mental Disorders

STUDY DESIGN:
Intervention Model Description: Participants are randomized either into a control group assigned to the standard of care diagnostic assessments once daily or into an experimental group assigned to the novel, personalized assessment system. The content of both assessment systems is the same, but the approach to delivering the assessments differs based on the arm. Each arm will have 25 participants, and any additional participants who register will be assigned to a waitlist.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All relevant participant research data is stored separate from protected health information and potentially identifiable information, including into which study arm the participant has been randomized.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Personalized, Transdiagnostic Assessments (Experimental): One or more times per day, participants in the Experimental Arm will be presented with a variable-length assessment based on the personalization algorithm. The assessment will include a dynamic number of questions based on personalized relevancy, engagement level, and assessment completion metrics. Questions are scored immediately upon submission, regardless of how many questions are answered. As questions are scored, the personalization algorithm takes the previous responses and response times into consideration when determining what and when to ask additional questions.
  Interventions: Diagnostic Test: Introspect Health
- Monotopic Assessments (Active Comparator): Once daily, participants in the Control Arm will be presented with the standard of care mental health surveillance assessments identified as relevant upon intake. The assessments will be scored in totality or not at all and have a fixed, predefined number of questions. No personalization of assessment will take place.
  Interventions: Diagnostic Test: Introspect Health

INTERVENTIONS:
Diagnostic Test: Introspect Health — Introspect Health is a software platform which has implemented both the monotopic and personalized, transdiagnostic assessment tools. The software is delivered via the internet using a mobile device or computer.

SUMMARY:
This study is investigating the self-report adherence and assessment completion rates when presented with a transdiagnostic, partial assessment multiple times a day when compared with a monotopic, complete assessment once a day. Specifically, the investigators are testing the hypothesis that the personalization of diagnostic assessment topics and timing will lead to improved self-report regiment adherence rates, assessment completion rates, and total assessments completed during the study period. The study does not test the efficacy of the personalized assessments as a diagnostic instrument, there is no clinical decision support provided to clinicians during this study, and there is no treatment provided during this study.

DETAILED DESCRIPTION:
Broadly, the goal of Introspect Health is to shift clinical practice from reactively treating psychiatric disorders and mental health issues once manifested to a preventative care model for integrative mental health in a way that is cost-effective and scalable. One of the principal areas of struggle in preventative mental health is self-report adherence and the ability for primary care physicians and non-psychiatrists to perform mental health surveillance with their patients. This study specifically examines the relationship between individuals and a novel self-report assessment tool. To do this, the investigators are performing a randomized controlled trial with two classes of users (the general public and patients undergoing treatment for mental health issues) for a six week trial comparing the novel self-report assessment tool to the standard of care assessment tools available to clinicians. Participants will be randomized to one of the two daily assessment regiments within the internet-delivered assessment tool: one that is representative of standard of care monitoring and one that is personalized both in terms of content and timing based on the participant's intake as well as ongoing participation. Neither the participants nor researcher will be aware of which arm the individual is randomized. After using the software for six weeks, the data will be analyzed specifically targeting self-adherence and assessment completion metrics to evaluate the potential benefits of a transdiagnostic assessment system over the standard-of-care monotopic assessment system. Assessment scoring is handled by an automated scoring engine, using the rules set forth by the standards in the assessment protocols. The study does not test the efficacy of the personalized assessments as a diagnostic instrument, there is no clinical decision support provided to clinicians during this study, and there is no treatment provided during this study.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* English fluency
* US citizen
* California resident
* Eligible to receive mental healthcare in the state of California
* Primary user of a smartphone device
* Daily access to Internet and email
* Meets a minimum level of 2.51 or higher on a self-rated technology use scale based on the average score of three Likert-style questions
* Willing to answer questions about themselves pertaining to physical and mental wellness throughout the Research Period

Exclusion Criteria:

* Undergoing care for condition requiring emergent treatment or hospitalization, including but not limited to: current or recent (within 3 months) acute manic or major depressive episode, clear and current suicidal risk, current or recent (within 3 months) history of substance abuse or drug dependence
* Undergoing active treatment for a condition wherein the additional burden of performing daily assessments may interfere with their pre-existing treatment regiment, cause undue anxiety, or risk inflammation of pre-existing issues
* Undergoing active treatment using a treatment modality that may adversely interact with research study participation such as psychopharmaceuticals affecting memory and cognition, therapeutic digital detox, or similar treatments
* Has ever participated in a Research Study testing the efficacy of transdiagnostic assessments, transdiagnostic interventions, or Internet-based CBT
* Additionally, patients on psychotropic medications are only eligible to be included while they maintain a stable dosage of their medication; if their medication dosage needs to change for any reason during the course of the Research Study, they would be required to withdraw from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-05 (Estimated); Primary Completion 2019-08 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
Self-Report Adherence Rate | 6 weeks
  Frequency of individuals adhering to the regiment of daily self-assessments, segmented by arm
Completed Assessments Scored | 6 weeks
  Total number of self-assessments completed throughout the study time frame, not including partial assessments, segmented by arm
Assessment Questions Scored | 6 weeks
  Total number of individual questions completed throughout the study time frame, segmented by arm

SECONDARY OUTCOMES:
Time per Assessment Question | 6 weeks
  Average time spent responding to each question during an assessment, segmented by arm and assessment
Response Time | 6 weeks
  Average time from initial assessment prompt to completion of the assessment, segmented by arm and assessment
Assessment Completion Rate | 6 weeks
  Frequency of individuals completing an assessment, segmented by arm and assessment

CONTACTS AND LOCATIONS:
Overall Officials: Anne M Huffman, PhD, Study Director — California Institute of Integral Studies; Michael K Owens, Principal Investigator — Introspect Health
Locations (1):
- California Institute of Integral Studies, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No
No IPD will be released. Statistical analysis of masked participant data will be published alongside one or more reports.